CLINICAL TRIAL: NCT03069040
Title: The Randomized Controlled Trial of Nerve Sparing Hysterectomy Radical Hysterectomy and Radical Hysterectomy
Brief Title: Nerve Sparing Radical Hysterectomy VS Radical Hysterectomy: Safety and Clinical Efficacy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Chen Chunlin (Other)
Responsible Party: Sponsor-Investigator, Chen Chunlin, Obstetrics and Gynecology, Southern Medical University, China
Organization: Southern Medical University, China (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SNSRH001
Record Dates: First submitted 2017-02-27; First posted 2017-03-03 (Actual); Last update posted 2017-03-03 (Actual); Status verified 2017-02

CONDITIONS: Cervical Cancer
Keywords: cervical cancer; NSRH; RH; urine flow mechanics; anorectal dynamics
MeSH Terms: conditions — Uterine Cervical Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- nerve-sparing radical hysterectomy (Experimental): The patient recived surgury of nerve-sparing radical hysterectomy.
  Interventions: Procedure: nerve sparing radical hysterectomy
- radical hysterectomy (Active Comparator): The patient recived surgury of radical hysterectomy.
  Interventions: Procedure: radical hysterectomy

INTERVENTIONS:
Procedure: nerve sparing radical hysterectomy — Type C1 radical hysterectomy,that is nerve sparing radical hysterectomy, requires separation of two parts of the dorsal parametria: the medialpart , which entails recto -uterineandrecto-vaginal ligaments, and the lateral laminar structure, also called mesoureter, which contains the hypogastric plexus. Furthermore, type C1 requires only a partial dissection of the ureter from the ventral parametria, which is usually asymmetric towards more extensive resection of the medial leaf of the cranial (above the ureter) part of the ventral parametria .
  Other Names: Type C1 radical hysterectomy
  Arms: nerve-sparing radical hysterectomy
Procedure: radical hysterectomy — In the C2 type, the ureter is completely dissected from the ventral parametria up to the urinary bladder wall. Defining the resection limits on the longitudinal (deep parametrial or vertical) plane is crucial for distinguishing between types C1 and C2.
  Other Names: Type C2 radical hysterectomy
  Arms: radical hysterectomy

SUMMARY:
Cervical cancer in young patients increased significantly in recent years, and early surgical treatment for patients with 5 years of survival rate is as high as 90%, But the traditional extensive hysterectomy (RH) caused by intraoperative pelvic autonomic nerve may damage the bladder and rectum and the incidence of complications such as sexual dysfunction is nearly 25% to 80%, thus seriously affect the patient's quality of life.Pelvic autonomic nerve preservation system of extensive hysterectomy (NSRH) can decrease the complications of above, but at home and abroad mainly adopts pulling the urine tube time, determination methods of residual urine volume, bladder function are studied in only a few scholars urine flow mechanics method is applied to carry on objective appraisal limited cases of postoperative bladder function, and the anorectal function damage ，we can use the anorectal dynamics to get objective index of anorectal function .overall research lack of large sample research of dynamic system. No objective index to evaluate the anorectal function In the early stage of the study, we have conducted about uterine ligament, sacral ligaments and nerve distribution of the bladder cervix vaginal ligament of experimental research, provide the neural anatomy basis for NSRH operation, and based on research for innovative operation scheme is put forward.Proposed on the basis of the above research, this study adopt the internationally used - urine flow mechanics, the method for evaluating the bladder function of NSRH, RH, two kinds of the injured function of bladder surgery patients before and after operation of comparative study, the change of dynamic assessment before and after surgery in patients with bladder function,and the anorectal function dameage and than provide the basis for further treatment.

ELIGIBILITY:
Inclusion Criteria:

* Cervical Cancer FIGO(2009) IA2,IB1,IB2,IIA1,IIA2

Exclusion Criteria:

* Cervical Cancer FIGO(2009) > IIb
* Patients received radiotherapy before opration
* The patient refused to sign a consent form.

Ages: 20 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2011-11-01 (Actual); Primary Completion 2017-12-31 (Estimated); Study Completion 2017-12-31 (Estimated)

PRIMARY OUTCOMES:
Survival rates | 5 years after operation
  Live or die
The recurrence rate | 5 years after operation
  Whether the tumor recurrence
Abdominal pressure urination | 1 years after operation
  Urine flow dynamic test results

SECONDARY OUTCOMES:
Abdominal pressure urination | 3 months after operation
  Urine flow dynamic test results
Abdominal pressure urination | 6 months after operation
  Urine flow dynamic test results
the results of anorectal dynamics | 1 months after opration
  the results of anorectal dynamics
the results of anorectal dynamics | 3 months after opration
  the results of anorectal dynamics
the results of anorectal dynamics | 6 months after opration
  the results of anorectal dynamics

CONTACTS AND LOCATIONS:
Locations (1):
- Southern Medical Universtity, China, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No